CLINICAL TRIAL: NCT02595814
Title: International Registry to Assess mEdical Practice With lOngitudinal obseRvation for Treatment of Heart Failure
Brief Title: Global Non-interventional Heart Failure Disease Registry
Acronym: REPORT-HF
Status: Terminated | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRPORTHF
Record Dates: First submitted 2015-10-13; First posted 2015-11-03 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Acute Heart Failure
Keywords: Registry; Heart failure; Hospitalized; Global; Morbidity; Mortality; Quality of life; AHF
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The clinical characteristics, initial presentation, management, and outcomes of patients hospitalized with new-onset (first diagnosis) heart failure (HF) or decompensation of chronic HF are poorly understood worldwide. REPORT-HF is a global, prospective, and observational HF disease registry designed to characterize patient trajectories longitudinally during and following an index hospitalization for acute HF.

ELIGIBILITY:
Inclusion Criteria:

Patients at least 18 years old, or older for those countries where the adult age is above 18 years of age, hospitalized with a primary diagnosis of acute heart failure.

Exclusion Criteria:

1-Concomitant participation in any/a clinical trial with any investigational treatment (for any sponsor).

2. Use of investigational drugs within 5 half-lives of enrollment, or until the expected pharmacodynamic effect has returned to baseline, whichever is longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollment of adult patients hospitalized with a primary diagnosis of acute Heart Failure (HF), i.e. new-onset (first diagnosis) HF or decompensation of chronic HF
Sampling Method: Probability Sample
Enrollment: 18805 (Actual)
Dates: Start 2014-07-23 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with different characteristics of heart faliure (HF) at hospitalization | From admission to discharge of the patient's index hospitalization (minimum 24 hours)
Percentage of patients who die during the index hospitalization | From admission to discharge of the patient's index hospitalization (minimum 24 hours)
Percentage of patients who die during the follow-up period post-discharge | up to 3 years
Percentage of patients who are re-hospitalized by primary re-hospitalization reason (Cardiovascular and non-Cardiovascular) | up to 3 years
Number of patients with different characteristics of post-discharge patient management | up to 3 years
Healthcare Resource Utilization assessed by number of patients with re-hospitalizations | up to 3 years

SECONDARY OUTCOMES:
Health-related Quality of life (HRQoL) based on patient reported data as measured by EQ-5D and the Kansas City Cardiomyopathy Questionnaire (KCCQ) questionnaires | up to 3 years
Caregiver burden based on Caregiver Burden Questionnaire -Heart Failure (CBQ-HF) and Work Productivity and Activity Impairment (WPAI) questionnaires | up to 3 years
Correlation ratio between practice patterns and outcomes | up to 3 years

CONTACTS AND LOCATIONS:
Locations (280):
- United States (13):
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Stony Brook, New York
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
- Algeria (2):
  - Novartis Investigative Site, Algiers
  - Novartis Investigative Site, Oran
- Argentina (10):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires, Buenos Aires F.D.
  - Novartis Investigative Site, Coronel Suarez, Buenos Aires F.D.
  - Novartis Investigative Site, Resistencia, Chaco Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Corrientes
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Mendoza
  - Novartis Investigative Site, Salta
- Australia (4):
  - Novartis Investigative Site, Gosford, New South Wales
  - Novartis Investigative Site, Auchenflower, Queensland
  - Novartis Investigative Site, Greenslopes, Queensland
  - Novartis Investigative Site, Bedford Park
- Austria (4):
  - Novartis Investigative Site, Eisenstadt
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Mödling
  - Novartis Investigative Site, Vienna
- Brazil (10):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, Tatuí, São Paulo
  - Novartis Investigative Site, Curitiba
  - Novartis Investigative Site, Recife
  - Novartis Investigative Site, Rio de Janeiro
  - Novartis Investigative Site, Sao Jose Do Rico Preto
- Bulgaria (4):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Canada (5):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Sainte-Foy, Quebec
- Chile (3):
  - Novartis Investigative Site, San Miguel, Santiago Metropolitan
  - Novartis Investigative Site, Concepción
  - Novartis Investigative Site, Santiago
- China (21):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Fuzhou, Fujian
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Baotou, Inner Mongolia
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Dalian, Liaoning
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Hangzhou
  - Novartis Investigative Site, Jinan
  - Novartis Investigative Site, Luoyang
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Taiyuan
  - Novartis Investigative Site, Ürümqi
  - Novartis Investigative Site, Wuhan
  - Novartis Investigative Site, Xiamen
  - Novartis Investigative Site, Yangzhou
  - Novartis Investigative Site, Zhengzhou
- Colombia (7):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Bogotá, Cundinamarca
  - Novartis Investigative Site, Bucaramanga, Santander Department
  - Novartis Investigative Site, Armenia
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Cali
- Ecuador (4):
  - Novartis Investigative Site, Guayaquil, Guayas
  - Novartis Investigative Site, Quito, Pichincha
  - Novartis Investigative Site, Guayaquil
  - Novartis Investigative Site, Portoviejo
- Egypt (4):
  - Novartis Investigative Site, Alexandria
  - Novartis Investigative Site, Cairo
  - Novartis Investigative Site, El Menia, Upper Egypt
  - Novartis Investigative Site, Suez Canal Region
- Germany (13):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Würzburg
- Greece (7):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Glyfada
  - Novartis Investigative Site, Ioannina
  - Novartis Investigative Site, Piraeus
  - Novartis Investigative Site, Thessaloniki
- Novartis Investigative Site, Guatemala City, Guatemala
- India (17):
  - Novartis Investigative Site, Panjim, Goa
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Vadodara, Gujarat
  - Novartis Investigative Site, Gurgaon, Haryana
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Manipal, Karnataka
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Amritsar, Punjab
  - Novartis Investigative Site, Ludhiana, Punjab
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, India
  - Novartis Investigative Site, Mumbai
  - Novartis Investigative Site, New Delhi
- Indonesia (9):
  - Novartis Investigative Site, Tangerang, Banten
  - Novartis Investigative Site, East Jakarta, DKI Jakarta
  - Novartis Investigative Site, South Jakarta, DKI Jakarta
  - Novartis Investigative Site, West Jakarta, DKI Jakarta
  - Novartis Investigative Site, Surabaya, East Java
  - Novartis Investigative Site, Medan, North Sumatera
  - Novartis Investigative Site, Bandung, West Java
  - Novartis Investigative Site, Bekasi, West Java
  - Novartis Investigative Site, Padang, West Sumatra
- Israel (4):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Nazareth
  - Novartis Investigative Site, Sefad
- Japan (7):
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Kure, Hiroshima
  - Novartis Investigative Site, Sakaidechō, Kagawa-ken
  - Novartis Investigative Site, Kita-ku, Okayama-ken
  - Novartis Investigative Site, Hirakata, Osaka
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Nagasaki
- Jordan (2):
  - Novartis Investigative Site, Amman
  - Novartis Investigative Site, Irbid
- Lebanon (4):
  - Novartis Investigative Site, El Chouf, LBN
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, Byblos
  - Novartis Investigative Site, Saida
- Malaysia (5):
  - Novartis Investigative Site, Alor Star, Kedah
  - Novartis Investigative Site, Kota Bharu, Kelantan
  - Novartis Investigative Site, Pulau Pinang, Pulau Pinang
  - Novartis Investigative Site, Johor Bahru
  - Novartis Investigative Site, Kuala Lumpur
- Mexico (5):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Culiacán, Sinaloa SN
  - Novartis Investigative Site, Aguascalientes
  - Novartis Investigative Site, San Luis Potosí City
  - Novartis Investigative Site, Xalapa
- Morocco (3):
  - Novartis Investigative Site, Casablanca
  - Novartis Investigative Site, Marrakesh
  - Novartis Investigative Site, Rabat
- Netherlands (6):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Leiderdorp
  - Novartis Investigative Site, Sneek
  - Novartis Investigative Site, Venlo
  - Novartis Investigative Site, Zwolle
- Norway (3):
  - Novartis Investigative Site, Hønefoss
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Skien
- Panama (2):
  - Novartis Investigative Site, San Jose de David, Provincia de Panamá
  - Novartis Investigative Site, Panama City
- Philippines (7):
  - Novartis Investigative Site, Baguio City, Baguio
  - Novartis Investigative Site, Cagayan de Oro City, Cagayan Valley
  - Novartis Investigative Site, Cebu City, Cebu
  - Novartis Investigative Site, Davao City, Davao Region
  - Novartis Investigative Site, Quezon City, Manila
  - Novartis Investigative Site, Manila, National Capital Region
  - Novartis Investigative Site, Angeles City, Pampanga
- Romania (7):
  - Novartis Investigative Site, Cluj-Napoca, Napoca
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Buzău
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Focşani
  - Novartis Investigative Site, Lasi
  - Novartis Investigative Site, Timișoara
- Russia (14):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, S-Petersburg
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Stavropol
  - Novartis Investigative Site, Tyumen
  - Novartis Investigative Site, Ulyanovsk
  - Novartis Investigative Site, Vladivostok
  - Novartis Investigative Site, Volgograd
- Saudi Arabia (4):
  - Novartis Investigative Site, Al Ahsa
  - Novartis Investigative Site, Dammam
  - Novartis Investigative Site, Khamis Mushait
  - Novartis Investigative Site, Riyadh
- South Africa (4):
  - Novartis Investigative Site, Durban, KwaZulu-Natal
  - Novartis Investigative Site, Bloemfontein
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Rivonia
- South Korea (10):
  - Novartis Investigative Site, Gyeonggi-do, Bucheon-si
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Daejeon, Korea
  - Novartis Investigative Site, Cheongju-si, North Chungcheong
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Pusan
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Suwon
  - Novartis Investigative Site, Taegu
- Spain (12):
  - Novartis Investigative Site, Mallorca, Balearic Islands
  - Novartis Investigative Site, Barakaldo, Basque Country
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Tarragona, Catalonia
  - Novartis Investigative Site, Mérida, Extremadura
  - Novartis Investigative Site, Las Palmas de Gran Canaria, Las Palmas de G.C
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, León
  - Novartis Investigative Site, Murcia
- Sweden (6):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Helsingborg
  - Novartis Investigative Site, Karlshamn
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Trollhättan
- Switzerland (3):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bruderholz
  - Novartis Investigative Site, Zurich
- Taiwan (4):
  - Novartis Investigative Site, Linkou District
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
- Thailand (5):
  - Novartis Investigative Site, Muang, Muang
  - Novartis Investigative Site, Muang, Thailand
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Tunisia (3):
  - Novartis Investigative Site, Monastir
  - Novartis Investigative Site, Sousse
  - Novartis Investigative Site, Tunis
- Turkey (Türkiye) (8):
  - Novartis Investigative Site, Pendik / Istanbul, Turkey
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Bursa
  - Novartis Investigative Site, Diskapi / Ankara
  - Novartis Investigative Site, Haydarpasa/Istanbul
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Meselik / Eskisehir
  - Novartis Investigative Site, Sivas
- United Arab Emirates (3):
  - Novartis Investigative Site, Abu Dhabi
  - Novartis Investigative Site, Al Ain City
  - Novartis Investigative Site, Dubai
- United Kingdom (10):
  - Novartis Investigative Site, Edgbaston, Birmingham
  - Novartis Investigative Site, Stockton-on-Tees, Cleveland
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Chesterfield, Yorkshire
  - Novartis Investigative Site, Herts, Yorkshire
  - Novartis Investigative Site, Chesterfield
  - Novartis Investigative Site, Telford
  - Novartis Investigative Site, Uxbridge
  - Novartis Investigative Site, Wakefield
  - Novartis Investigative Site, York
- Novartis Investigative Site, Ho Chi Minh City, Vietnam

REFERENCES:
- [Background] Filippatos G, Khan SS, Ambrosy AP, Cleland JG, Collins SP, Lam CS, Angermann CE, Ertl G, Dahlstrom U, Hu D, Dickstein K, Perrone SV, Ghadanfar M, Bermann G, Noe A, Schweizer A, Maier T, Gheorghiade M. International REgistry to assess medical Practice with lOngitudinal obseRvation for Treatment of Heart Failure (REPORT-HF): rationale for and design of a global registry. Eur J Heart Fail. 2015 May;17(5):527-33. doi: 10.1002/ejhf.262. Epub 2015 Mar 10. PMID 25754836
- [Derived] Tay WT, Teng TK, Ouwerkerk W, Cleland JGF, Collins SP, Angermann CE, Dickstein K, Dahlstrom U, Schweizer A, Obergfell A, Yiu KH, Ghadanfar M, Hassanein M, Ren QW, Gu WL, Ertl G, Perrone SV, Filippatos G, Lam CSP, Tromp J. Global patterns of polypharmacy after acute heart failure hospitalization: Prevalence and outcomes from the REPORT-HF registry. Eur J Heart Fail. 2025 Oct 1. doi: 10.1002/ejhf.70056. Online ahead of print. PMID 41031485
- [Derived] Chyou JY, Tay WT, Tromp J, Ouwerkerk W, Yiu KH, Cleland JGF, Collins SP, Angermann CE, Ertl G, Dahlstrom U, Dickstein K, Perrone SV, Ghadanfar M, Schweizer A, Obergfell A, Filippatos G, Lam CSP. Prognostic Implications and Global Perspectives of Atrial Fibrillation in Patients Hospitalized for Heart Failure. JACC Heart Fail. 2025 Mar;13(3):453-464. doi: 10.1016/j.jchf.2024.11.009. Epub 2025 Feb 5. PMID 39918534
- [Derived] Ouwerkerk W, Tromp J, Cleland JGF, Angermann CE, Dahlstrom U, Ertl G, Hassanein M, Perrone SV, Ghadanfar M, Schweizer A, Obergfell A, Dickstein K, Filippatos G, Collins SP, Lam CSP. Association of time-to-intravenous furosemide with mortality in acute heart failure: data from REPORT-HF. Eur J Heart Fail. 2023 Jan;25(1):43-51. doi: 10.1002/ejhf.2708. Epub 2022 Nov 23. PMID 36196060